CLINICAL TRIAL: NCT05698966
Title: Low Dose Antenatal Corticosteroids for Late Preterm Delivery (LoDAC Study)
Brief Title: Low Dose Antenatal Corticosteroids for Late Preterm Delivery
Acronym: LoDAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ron Beloosesky MD, Head of ultrasound in obstetrics and gynecology, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00451890
Record Dates: First submitted 2022-12-31; First posted 2023-01-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Morbidity; Preterm Labor
Keywords: corticosteroids; low dose; late prerterm
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- betamethasone 12 mg (Active Comparator): 3 mg betamethasone sodium phosphate and 3 mg betamethasone acetate per milliliter. The first dose of study drug medication will be administered at randomization as 2 ml injection; the next dose of 2 ml will be administered 24 hours later
  Interventions: Other: we will use reduced dose of acceptable corticosteroids treatment for preterm birth
- betamethasone 3 mg (Experimental): 3 mg betamethasone sodium phosphate and 3 mg betamethasone acetate per milliliter. The first dose of study drug medication will be administered at randomization as 0.5 ml injection; the next dose of 0.5 ml will be administered 24 hours later
  Interventions: Other: we will use reduced dose of acceptable corticosteroids treatment for preterm birth

INTERVENTIONS:
Other: we will use reduced dose of acceptable corticosteroids treatment for preterm birth — the two different group will differ in the doses of corticosteroids

SUMMARY:
This is a study proposal for a clinical trial to evaluate the effectiveness of a reduced dose of antenatal betamethasone (a steroid medication) in preventing respiratory problems in late preterm infants (born between 34 and 36 weeks of gestation). The study will be conducted in medical centers in Israel and will involve women who are at high risk for delivering a late preterm infant. The participants will be randomly assigned to receive either a full dose (12 mg) or a quarter dose (3 mg) of betamethasone, administered 24 hours apart. The main outcome measure of the study will be the incidence of respiratory problems or neonatal death within 72 hours of delivery in the two groups. The study is designed to determine if the reduced dose of betamethasone is non-inferior (i.e., not significantly worse) than the full dose in preventing respiratory problems in late preterm infants.

DETAILED DESCRIPTION:
Antenatal corticosteroids (ACS) are a type of steroid medication that is administered to pregnant women at risk of preterm birth in order to reduce the risk of respiratory distress syndrome (RDS) and other complications in the newborn. ACS were first demonstrated to be effective in a controlled trial conducted in the 1970s by Liggins and Howie, who used a combination of betamethasone at a dose of 12 mg given in two doses 24 hours apart. Since then, numerous randomized controlled trials and meta-analyses have shown that ACS can significantly reduce neonatal death, RDS, intraventricular hemorrhage, necrotizing enterocolitis, and the need for respiratory support and neonatal intensive care unit admission in preterm infants. ACS are now recommended for use in virtually all pregnancies at risk of preterm delivery between 24 and 34 weeks of gestation. The use of ACS in late preterm pregnancies (between 34 and 37 weeks) has also been studied, with mixed results. The largest study to date, the ALPS trial, found that ACS reduced composite adverse outcomes and respiratory morbidity in late preterm infants, but did not significantly reduce the risk of RDS or mortality. The American Congress of Obstetricians and Gynecologists has recommended the use of ACS in late preterm pregnancies, but with caution due to the potential for adverse effects such as hypoglycemia. Long-term follow-up studies are needed to evaluate the potential long-term effects of ACS in late preterm infants. In this the participants will be randomly assigned to receive either a full dose (12 mg) or a quarter dose (3 mg) of betamethasone, administered 24 hours apart. The main outcome measure of the study will be the incidence of respiratory problems or neonatal death within 72 hours of delivery in the two groups. The study is designed to determine if the reduced dose of betamethasone is non-inferior (i.e., not significantly worse) than the full dose in preventing respiratory problems in late preterm infants.

ELIGIBILITY:
Inclusion Criteria:- - Singleton pregnancy at 34 weeks 0 days to 36 weeks 5 days of gestation at risk for / high probability of delivery in the late preterm period (34+0-36+5 weeks of gestation).

Criteria for determination of late preterm delivery risk:

1. Preterm uterine contractions with intact membranes, and at least 3 cm dilation or 75% cervical effacement
2. Spontaneous rupture of the membranes
3. Expected preterm delivery for any other indication via induction or cesarean between 24 hours to 7 days after the planned randomization, as determined by the obstetric provider.

   -

   Exclusion Criteria: They had already received a full course of betamethasone.
   * Expected delivery in less than 12 hours, irrespective of cause including: 1)ruptured membranes in the presence of more than 6 contractions per hour or cervical dilation of 3 centimeters or more unless oxytocin was withheld for at least 12 hours (although other induction agents were allowed), 2) chorioamnionitis, 3) cervical dilation of 8 cm or more, and 4) evidence of non-reassuring fetal status requiring immediate delivery.
   * Prior ACS treatment
   * Current known or suspected infection ( viral, bacterial or other)
   * Pre-gestational diabetes mellitus.
   * Any infection that required antibiotics or hospitalization in the month prior to study allocation - Poor understanding of the inform consent language

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1510 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory morbidity | first 72 hours after birth
  1. Use of continuous positive airway pressure (CPAP) or high-flow nasal cannula for ≥2 continuous hr in the first 72 hours
  2. Fraction of inspired oxygen of ≥0.30 for ≥4 continuous hr in the first 72 hours
  3. Mechanical ventilation in the firdt 72 hours yes/no
  4. extracorporeal membrane oxygenation (ECMO) yes/no
  5. TTN: transient tachypnea of newborn yes/no

SECONDARY OUTCOMES:
other neonatal morbidities other neonatal morbidities | first 30 days after birth
  for all the parameters: yes or no Severe respiratory complications (a composite outcome of CPAP or high-flow nasal cannula for at least 12 continuous hours, supplemental oxygen with a fraction of inspired oxygen of at least 0.30 for at least at least 24 continuous hours, ECMO or mechanical ventilation, stillbirth, or neonatal death within 72 hours after delivery) Respiratory distress syndrome, Transient tachypnea of the newborn, Apnea, Bronchopulmonary dysplasia, Surfactant administration, Need for resuscitation at birth , Feeding difficulty, Hypothermia, , Necrotizing enterocolitis, Intraventricular hemorrhage Papile grade 3 or 4, Neonatal sepsis, Pneumonia, Pulmonary air leak, Death before discharge
  Newborns blood levels of glucose: mg/dl insulin and c-peptide : levels in serum

CONTACTS AND LOCATIONS:
Locations (16):
- Israel (16):
  - Emek Medical Center, Afula
  - Kaplan Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Hilel Yafee Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rambam Health Care Cmpus, Haifa
  - Hadassah Ein Karem, Jerusalem
  - Hadassah Har Hzofim, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir medical center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided